CLINICAL TRIAL: NCT00788762
Title: Myocilin Variations and Familial Glaucoma in Taxiarchis, A Small Greek Village.
Brief Title: Myocilin Variations and Familial Glaucoma in Taxiarchis
Acronym: Taxiarchis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Other Study IDs: A6798
Record Dates: First submitted 2008-11-07; First posted 2008-11-11 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Glaucoma
Keywords: glaucoma; myocilin
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Myocilin screening was performed from blood or saliva specimens taken from the village. The promoter region and exons 1-3 of myocilin were sequenced at the Portland Veterans Administration Medical center. Microsatellite marker analysis in the GLC1A region, including D1S452, D1S1619, D1S2790 and D1S242 was performed at deCODE (Reykjavik, Iceland).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Villagers in Taxiarchis

SUMMARY:
Taxiarchis, a small village in Northern Greece with 1060 inhabitants, was considered to have a surprisingly high incidence of glaucoma. This isolated population located on Mount Holomondas appeared to be enriched for familial glaucoma. Based upon the high reported incidence of glaucoma in Taxiarchis and previous findings of the Thr377Met myocilin mutation in the Greek population,the investigators undertook a community-based study to determine if this variant was present in this village.

ELIGIBILITY:
Inclusion Criteria:

* Individuals born in Taxiarchis

Exclusion Criteria:

* Individuals that have not been born in Taxiarchis

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Villagers from Taxiarchis
Sampling Method: Non-Probability Sample
Enrollment: 840 (Estimated)
Dates: Start 2007-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Examining all of the villagers to determine the actual incidence of glaucoma in Taxiarchis and identify the Thr377Met myocilin mutation in glaucoma patients. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Anastasios G Konstas, MD, PhD, Principal Investigator — Glaucoma Unit, 1st University Dept
Locations (1):
- Taxiarchis village, Polygyros, Halkidiki, Greece